CLINICAL TRIAL: NCT03163225
Title: Characterizing and Quantifying Challenges and Opportunities in Outpatient Care
Brief Title: Opportunities in Outpatient Care
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050460
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Outpatient Care
Keywords: outpatient care; emergency department visits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study is to determine whether there are things that Intermountain can do to break down barriers to helping patients see their primary doctors or other outpatient clinics. To do this we will develop and test a classification scheme to help us understand how we might reduce some avoidable emergency department and InstaCare visits.

DETAILED DESCRIPTION:
The study will develop a first-pass taxonomy that classifies the causes and effects of challenges and opportunities of outpatient care leading to potentially avoidable ED and urgent care center visits.

The study will quantify the proportion of ED and urgent care center visits that result from a challenge or opportunity in outpatient care and classify the causes and outcomes according to the taxonomy. It will also define the 30 and 90 day episode costs of ED and urgent care center visits associated with a challenges and opportunities of outpatient care beginning the day of the ED or urgent care center visit.

ELIGIBILITY:
Inclusion Criteria:

* All Emergency Department/IC patients who can consent, including children.

Exclusion Criteria:

* Unable to give consent
* Prisoners

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department/InstaCare patients
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of avoidable ED visits due to a "missed" opportunity in outpatient care | 1 Day
  The proportion of ED visits during the selected shifts that were deemed to be potentially avoidable according to the developed taxonomy
Incidence rate of avoidable InstaCare visits due to a "missed" opportunity in outpatient care | 1 Day
  The proportion of Instacare visits during the selected shifts that were deemed to be potentially avoidable according to the developed taxonomy

SECONDARY OUTCOMES:
Patient Disposition Status from the ED | 1 Day
  Disposition status from after the ED visit, collected from the medical record. Status will be one of the following: admitted, observation, transfer to facility, discharged, deceased.
Patient Disposition Status from the InstaCare | 1 Day
  Disposition status from after the Instacare visit, collected from the medical record. Status may be admitted, observation, transfer to facility, discharged, or deceased.
Length of stay for admitted patients | Up to 30 days
  Length in stay by days in study patients admitted to the hospital
Harms to patients due to the missed opportunities in outpatient care. | 90 days
  Categorization of the "harms" on patients due to the missed opportunities in outpatient care using NCC-MERP categorizations
30 day episode costs | 30 days
  All attributable healthcare costs accrued to study patients from the date of visit to +30 days.
90 day episode costs | 90 days
  All attributable healthcare costs accrued to study patients from the date of visit to +90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Allen, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (9):
- United States (9):
  - Cottonwood InstaCare, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - Riverton Hospital, Riverton, Utah
  - Southridge InstaCare, Riverton, Utah
  - Salt Lake City InstaCare, Salt Lake City, Utah
  - Memorial InstaCare, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Sandy InstaCare, Sandy City, Utah
  - Alta View Hospital, Sandy City, Utah

IPD SHARING:
Plan to Share IPD: No